CLINICAL TRIAL: NCT06573541
Title: Use of Ultrasound in the Initial Management of Patients in Shock in the Nancy Emergency Department - Retrospective Descriptive Analysis
Brief Title: Use of Ultrasound in the Initial Management of Patients in Shock in the Nancy Emergency Department
Status: Active, not recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, HUOT-MARCHAND Matthieu, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2024-A01851-46
Record Dates: First submitted 2024-08-19; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Shock
Keywords: shock; ultrasound; emergency department
MeSH Terms: conditions — Shock; Emergencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group receiving ultrasound
  Interventions: Device: Use of ultrasound
- group not receiving ultrasound

INTERVENTIONS:
Device: Use of ultrasound — Use of ultrasound in the initial management of patients in shock
  Groups: group receiving ultrasound

SUMMARY:
Context: shock is a serious pathology where diagnostic and therapeutic speed determines the prognosis, ultrasound can be a valuable aid for the emergency physician to differentiate the different types of shock and allow appropriate treatment.

Hypothesis: what are the uses of ultrasound in the initial diagnostic and therapeutic management of patients in shock at the Emergency Department of Nancy? Main outcome: Describe the use of ultrasound in the initial diagnostic and therapeutic management of patients in shock at the Nancy Emergency Department Secondary outcome: Study the contribution of the use of different ultrasound techniques in the initial diagnostic and therapeutic management of patients depending on the type of shock state

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Shock (MAP < 65 mmHg + lactate ≥ 2 mmol/l)
* Admission to the Nancy ED between 01/01/2023 and 12/31/2023
* ICD-10 output coding: R57: shock, not elsewhere classified; R570: cardiogenic shock; R571: hypovolemic shock; R572: septic shock; R578: other shocks; R579: shock, unspecified; T794: traumatic shock; T782: anaphylactic shock, unspecified; or diagnosis of entry into intensive care including the word "shock"

Exclusion Criteria:

* Age < 18 years old
* Absence of shock
* No passage through the Nancy ED
* Patient whose initial treatment was carried out in another emergency department
* State of shock occurring after going to the emergency department

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults in shock at the Nancy ED
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
rate of ultrasound use | Day 0
  use of different types of ultrasound or not for diagnostic and therapeutic purposes depending on the type of shock state

SECONDARY OUTCOMES:
rate of patients with care changes | Day 0
  changes in initial diagnostic and therapeutic management when an ultrasound technique is used compared to patients who did not benefit from it (duration of passage to ED and treatment, time until diagnosis, vascular filling rate, catecholamine utilization rate)

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU, Nancy, France

IPD SHARING:
Plan to Share IPD: No